CLINICAL TRIAL: NCT07040371
Title: A Health Promotion Behavior Intervention for Elderly Migrants: a Randomized Controlled Trial
Brief Title: Health Promotion Behavior Intervention for Elderly Migrants to Improve Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huzhou University (Other)
Responsible Party: Principal Investigator, Li Fang, Principal Investigator, Huzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 202401-36
Record Dates: First submitted 2025-06-25; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Elderly Migrants; Health Promotion Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Promotion Behavior Intervention + Routine Community Nursing and Management (Experimental): In addition to routine community nursing and management, the experimental group of elderly migrants also received the health promotion behavior intervention program developed in this study.
  Interventions: Other: Health Promotion Behavior Intervention Program
- routine community nursing and management only (Active Comparator): The control group of elderly migrants received routine community nursing and management, which primarily included distributing health manuals, conducting regular health education activities, follow-up visits, etc.
  Interventions: Other: receiving routine community care and management only

INTERVENTIONS:
Other: Health Promotion Behavior Intervention Program — The intervention program is structured around a three-step framework: ① building motivation and providing opportunities; ② reinforcing motivation, enhancing capabilities, and providing opportunities; and ③ sustaining motivation, strengthening capabilities, and providing opportunities. The process involves assessing the current state of health-promoting behaviors among elderly migrants, implementing interventions to promote these behaviors, and evaluating the effectiveness of the interventions. The program spans 12 weeks and is carried out by a team of researchers and nursing students. Key intervention components include: ① helping elderly migrants recognize their health issues, analyzing the impact of migration on health-promoting behaviors, and emphasizing the importance of such behaviors through comparisons of negative and positive case studies; ② conducting thematic training on health habits, dietary nutrition, exercise safety, oral hygiene, and other topics through health lectures,
  Arms: Health Promotion Behavior Intervention + Routine Community Nursing and Management
Other: receiving routine community care and management only — It primarily included distributing health manuals, conducting regular health education sessions, and performing follow-ups. Researchers and community nurses collected and addressed health-related inquiries raised by the elderly migrants. Additionally, to ensure scientific rigor and equity in the study, compensatory interventions (such as providing equivalent intervention opportunities or distributing relevant intervention materials) were offered to participants based on their actual needs upon completion of the research project.
  Arms: routine community nursing and management only

SUMMARY:
This study aimed to develop a health promotion behavior intervention for elderly migrants and evaluate its effects, in order to provide insights for enhancing health-promoting behaviors among elderly migrants, improving community-based health management services for this population, and addressing health challenges related to migration in an aging society.

DETAILED DESCRIPTION:
This study employed a randomized controlled trial design, with elderly migrants in Huzhou City as participants, randomly assigned to either an intervention or control group. The control group received routine community care, while the intervention group underwent a 12-week "Health Promotion Behavior Intervention Program for Elderly Migrants" based on the Behaviour Change Wheel (BCW) theory. The intervention targeted motivation, capability, and opportunity through six dimensions, including health habits, social participation, and health responsibility, delivered via group interactions, face-to-face sessions, online resources, and community activities. Standardized scales were used to assess health promotion behaviors, self-perceived aging, family care, and loneliness at baseline, 6 weeks, and post-intervention. Data analysis involved Shapiro-Wilk tests, Mann-Whitney U tests, and Wilcoxon signed-rank tests.

ELIGIBILITY:
Inclusion Criteria:

* Age requirement: female ≥55 years, male ≥60 years；
* Residing in Huzhou city for >6 months;
* Voluntary participation with signed informed consent;
* Cognitively intact.

Exclusion Criteria:

* Individuals with language/communication barriers.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
the geriatric health promotion scale | baseline, week 6, and week 12
  The health-promoting behaviors of elderly migrants were assessed using the the geriatric health promotion scale. This scale consists of 22 items across six dimensions: health habits, social participation, health responsibility, healthy diet, physical exercise, and oral health care. A 4-point Likert scale was used for scoring, with higher scores indicating better health-promoting behaviors. In this study, the Cronbach's α coefficient for this scale was 0.843, demonstrating good internal consistency reliability.

SECONDARY OUTCOMES:
the brief ageing perceptions questionnaire (B-APQ) | baseline, week 6, and week 12
  The Brief Ageing Perceptions Questionnaire (B-APQ) was used to assess self-perceptions of aging among elderly migrants. This 17-item scale evaluates five dimensions: timeline chronic, positive consequences, positive control, negative consequences, and emotional representations. Responses were scored using a 4-point Likert scale, with higher scores indicating more negative self-perceptions of aging. In the current study, the scale demonstrated acceptable internal consistency (Cronbach's α = 0.782).
The family APGAR | baseline, week 6, and week 12
  The family APGAR was employed to measure perceived family support among elderly migrants. This instrument assesses five domains: adaptability, partnership, growth, affection, and resolve, utilizing a 3-point Likert scale where higher scores indicate stronger family support. In the present study, the scale demonstrated excellent internal consistency with a Cronbach's α coefficient of 0.940.
UCLA Loneliness Scale | baseline, week 6, and week 12
  The UCLA Loneliness Scale (8-item version) was administered to evaluate loneliness levels among elderly migrants. This standardized instrument consists of 8 items rated on a 4-point Likert scale, with higher total scores indicating greater severity of loneliness. In the current study, the scale demonstrated good reliability (Cronbach's α = 0.841).

CONTACTS AND LOCATIONS:
Overall Officials: Meijuan Cao, Study Director — Huzhou University
Locations (1):
- Huzhou University, Huzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No